CLINICAL TRIAL: NCT07115667
Title: A Prospective Single-Arm Clinical Trial of Radiation Combined With BCMA/CD3 Bispecific Antibody Therapy for Solitary Bone Plasmacytoma With Mild Bone Marrow Infiltration
Brief Title: Radiation Combined With BCMA/CD3 Bispecific Antibody Therapy for Solitary Bone Plasmacytoma With Mild Bone Marrow Infiltration
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025065
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Solitary Bone Plasmacytoma; Plasmacytoma of Bone; Plasma Cell Disorders
Keywords: solitary bone plasmacytoma; BCMA/CD3 bispecific antibody

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BsAbs-treatment group (Experimental): Patients with solitary bone plasmacytoma (SBP) with mild bone marrow infiltration will receive radiation combined with a BCMA/CD3 bispecific antibody (CM336)
  Interventions: Drug: BCMA/CD3 bispecific antibody (CM336)

INTERVENTIONS:
Drug: BCMA/CD3 bispecific antibody (CM336) — Patients with solitary bone plasmacytoma (SBP) with mild bone marrow infiltration will receive radiation combined with a BCMA/CD3 bispecific antibody (CM336)

SUMMARY:
This is a prospective, single-arm, single-center clinical trial designed to evaluate the safety and efficacy of radiation combined with a BCMA/CD3 bispecific antibody (CM336) in patients with solitary bone plasmacytoma (SBP) with mild bone marrow infiltration.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center clinical trial designed to evaluate the safety and efficacy of radiation combined with a BCMA/CD3 bispecific antibody (CM336) in patients with solitary bone plasmacytoma (SBP) with mild bone marrow infiltration. SBP is a rare plasma cell malignancy with a high risk of progression to multiple myeloma (MM), particularly in patients with minimal bone marrow involvement.

Although radiotherapy is the standard treatment, it is often insufficient to eradicate clonal plasma cells and prevent progression in high-risk patients. CM336, a novel BCMA/CD3 bispecific antibody, has demonstrated promising activity in relapsed/refractory multiple myeloma. In this trial, eligible patients will receive radiotherapy followed by a 12-cycle limited treatment course of CM336, aiming to achieve deep clearance of residual malignant cells and reduce progression risk.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Histologically confirmed SBP with <10% clonal plasma cells in marrow
* ECOG ≤ 2
* No prior anti-myeloma therapy. Previous local radiotherapy for SBP is not an exclusion criterion.
* Meets laboratory and imaging criteria

Exclusion Criteria:

1. Patients who have previously received anti-plasma cell therapy, including melphalan, cyclophosphamide, proteasome inhibitors, immunomodulatory drugs, monoclonal antibodies, bispecific antibodies, or chimeric antigen receptor T-cell (CAR-T) therapy.
2. Any condition that, in the opinion of the investigator, would make the patient unsuitable for participation in this study.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | From first dose through 28 days after last dose
  The primary outcome is to evaluate the safety and tolerability of the combination therapy. This includes the incidence, severity, and type of adverse events (AEs) and serious adverse events (SAEs), graded according to NCI CTCAE v5.0. Particular attention will be paid to cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS). Safety assessments will include laboratory parameters, vital signs, ECGs, and clinical symptoms.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 5 years
  PFS is defined as the time from the start of treatment to the first documentation of disease progression or death from any cause, whichever occurs first. Disease progression will be assessed using IMWG criteria for progression from solitary plasmacytoma to multiple myeloma.
Multiple Myeloma Free Survival (MMFS) | Up to 5 years
  MMFS is defined as the time from the start of treatment to the first documented diagnosis of multiple myeloma, based on IMWG criteria. Patients who do not progress to MM will be censored at the date of last follow-up. The diagnosis of MM will be confirmed by clinical, laboratory, and imaging criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided